CLINICAL TRIAL: NCT03937180
Title: The Effectiveness of a Blended Care Program for the Discontinuation of Benzodiazepines Use for Sleeping Problems in Primary Care: a Clustered Randomized Trial.
Brief Title: Blended Care for the Discontinuation of Benzodiazepine Use
Acronym: Big Bird
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristien Coteur (Other)
Collaborators: Belgium Health Care Knowledge Centre (Other Government); Universiteit Antwerpen (Other); University Ghent (Other); Vrije Universiteit Brussel (Other); Université Libre de Bruxelles (Other); Université de Liège (Other)
Responsible Party: Sponsor-Investigator, Kristien Coteur, Project manager - p.p. Chief investigator prof. dr. Catharina Matheï, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S61194; KCE-17016 (Other Grant/Funding Number: KCE)
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Benzodiazepine Dependence; Benzodiazepine Dependent; Benzodiazepine Withdrawal
Keywords: benzodiazepines; blended care

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (Other): Patients will receive 'usual care' left at the discretion of the treating general practitioner (GP). They are expected to follow the Belgian guidelines, which propose education of the patient about the harmful effects of chronic benzodiazepines and z-drugs ((z-)BZD) use, the alternatives, and the advice to discontinue (z-)BZD use. A stepped approach is recommended. First, a minimal intervention strategy such as a discontinuation letter or a short advice is applied. If unsuccessful, a brief intervention, which may span one or more consults, is recommended. During such an intervention, the GP will - based on the principles of motivational interviewing- assess the patient's readiness for change and match the appropriate intervention. A tapering scheme will be developed which typically consists of a 10-20% reduction in the daily dose of the (z-)BZD every 2-4 weeks.
  Interventions: Behavioral: Usual care
- Blended care (Experimental): Usual care is supported by the use of an interactive e-tool. The e-tool provides psycho-education about sleep and sleep medication, and exercises featuring cognitive behavioural techniques to enhance the self-management of the patient. It's purpose is to motivate patients to discontinue the use of (z-)BZD, to adapt alternative remedies and to support them in this process. The patient can grant the participating GP access to all his answers in the e-tool, making it possible to discuss their findings and experiences face-to-face. During consultations, the GP will also assess the patients' readiness for change and match the appropriate intervention. A tailored gradual taper of the (z-)BZD will be agreed upon, which typically consists of a 10-20% reduction in the daily dose every 2-4 weeks. Follow-up appointments are scheduled depending on the needs of the patient until the end of dose reduction.
  Interventions: Behavioral: Blended care

INTERVENTIONS:
Behavioral: Blended care — An interactive e-learning programme delivered through a secured web-based platform for patients and general practitioners (GPs), blended with face-to-face contacts between the involved GP and patient.
  Arms: Blended care
Behavioral: Usual care — General practitioners offering usual care are expected to follow the Belgian guidelines as described in the most recent online version of "Anxiety, stress and sleeping problems A toolbox for general practitioners." or "Sleeping pills and sedatives. How to assist your patients in the search for other solutions?" which are both available in French and Dutch.
  Arms: Usual care

SUMMARY:
This study aims to compare two strategies performed by GPs to help patients taking benzodiazepines on a daily basis for at least six months to discontinue their use. The first strategy consists of the usual or standard support provided by the GP, which often starts with a discontinuation advice or letter, the second is blended support where face-to-face consultations with the GP are alternated with web-based self-learning by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and older capable of giving informed consent,
* Having his/her Global Medical File managed by one of the participating general practitioners
* Receiving prescriptions of (z-)BZDs from participating GP for use on a daily basis
* Reporting daily intake (≥ 80% of days) of (z-)BZDs in the last 6 months for a primary indication of sleeping problems

Exclusion Criteria:

* Presence of any severe psychiatric and neurologic condition that in the judgment of the treating GP implies a contraindication for (z-)BZD withdrawal
* Presence of terminal illness
* Any cases where stopping of (z-)BZDs might be harmful
* Unwillingness or inability to provide informed consent
* Not having e-literacy (being familiar with email and internet use)
* Patients with a substance use disorder (other than (z-)BZD) will also be excluded from the study because in these cases there is often a sub-therapeutic (z-)BZD dependence and/or comorbid psychological/psychiatric comorbid conditions requiring specialist care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 924 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that discontinued (z-)BZD use at 12 months assessed by toxicological screening | 12 months
  Long-term effect of a blended care approach versus usual care on the discontinuation of (z-)BZD

SECONDARY OUTCOMES:
Proportion of patients that discontinued (z-)BZD use at 6 months assessed by toxicological screening | 6 months
  Short-term effect of a blended care approach versus usual care on the discontinuation of (z-)BZD
EQ-5D-3L assessed at week 6, 12, 26 and 52 | 12 months
  Effect of a blended care approach versus usual care on the quality of life. The EQ-5D-3L is the three-level version of the EuroQol five dimension scale measuring quality of life.
Proportion of patients with self-reported discontinuation of (z-)BZD use assessed at week 6, 12, 26 and 52 | 12 months
  Effect of a blended care approach versus usual care on self-reported discontinuation of (z-)BZD use
The number of defined daily doses (DDD) of (z-)BZD prescribed in the preceding interval assessed at week 6, 12, 26 and 52 | 12 months
  Effect of a blended care approach versus usual care on the number of DDD of benzodiazepines prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Catharina Matheï, Study Chair — KU Leuven
Locations (110):
- Belgium (110):
  - Leysen Bert, Broechem, Antwerpen
  - Asselman Valerie, Hoboken, Antwerpen
  - Van Tongelen Sofie, Mechelen, Antwerpen
  - Thomas Pol, Jette, Brussels Capital
  - Maquet Elisabeth, Saint-Gilles, Brussels Capital
  - Fauquert Benjamin, Schaarbeek, Brussels Capital
  - Uhry Franck, Uccle, Brussels Capital
  - Vansintejan Johan, Vilvoorde, Brussels Capital
  - Bedoret Virginie, Woluwe-Saint-Pierre - Sint-Pieters-Woluwe, Brussels Capital
  - Catinus Pierric, Châtelineau, Henegouwen
  - Vanderstraeten Katrien, Berchem, Kluisbergen
  - Ceulemans Steven, Beverst, Limburg
  - Coolen Antoon, Beverst, Limburg
  - Geskens Valérie, Beverst, Limburg
  - Fransis Jan, Ham, Limburg
  - Stulens Jan, Hasselt, Limburg
  - Thys Eline, Hasselt, Limburg
  - Vernyns Sander, Hasselt, Limburg
  - Beenders Wim, Maaseik, Limburg
  - Vanleeuw Ben, Zolder, Limburg
  - Kang Thida, Boncelles, Luik
  - Deleu Gabriel, Hodeige, Luik
  - Andre Jean-François, Liège, Luik
  - Rousseau Cecile, Liège, Luik
  - Steyaert Elodie, Neupré, Luik
  - Debry Jean-Yves, Ougrée, Luik
  - Evrard Antoine, Tilff, Luik
  - Parada Alberto, Trois-Ponts, Luik
  - Cohnen Ingrid, Waimes, Luik
  - Germay Arlette, Libin, Luxemburg
  - Gueibe France, Libin, Luxemburg
  - De Vleeschouwer Oriane, Saint-Hubert, Luxemburg
  - Vanschepdael Céline, Saint-Hubert, Luxemburg
  - Mattart Jacques, Andenne, Namen
  - Lafontaine Jean Baptiste, Namur, Namen
  - Kerckvoorde Lien, Aalter, Oost-Vlaanderen
  - Mahieu Inge, Asper, Oost-Vlaanderen
  - Cuelenaere Maarten, Assenede, Oost-Vlaanderen
  - De Sadeleer Jo, Borsbeke, Oost-Vlaanderen
  - Degrave Stijn, Herzele, Oost-Vlaanderen
  - De Muynck Kim, Kaprijke, Oost-Vlaanderen
  - Van Marcke Maarten, Lebbeke, Oost-Vlaanderen
  - Joos Ellen, Nevele, Oost-Vlaanderen
  - Everaert Leen, Nevele, Oost-Vlaanderen
  - Vermeulen Sofie, Sint-Martens-Latem, Oost-Vlaanderen
  - Heyerick Maaike, Zulte, Oost-Vlaanderen
  - Lemlijn Nathalie, Kessel-Lo, Vlaams-Brabant
  - Heijmans Stephane, Linkebeek, Vlaams-Brabant
  - Pening Maud, Nivelles, Waals-Brabant
  - Lens Marie, Ottignies, Waals-Brabant
  - Massaux Godelieve, Wavre, Waals-Brabant
  - De Vlieghere Marieke, Jabbeke, West-Vlaanderen
  - Caenepeel Laurens, Koksijde, West-Vlaanderen
  - Delvaux Nicolas, Lissewege, West-Vlaanderen
  - Knockaert Iris, Lissewege, West-Vlaanderen
  - Demeyere Tijs, Moorslede, West-Vlaanderen
  - Vandenameele Steffi, Sijsele, West-Vlaanderen
  - De Sutter Inge, Aalst
  - Maenen Arjen, Alken
  - Janssen Marie-Eve, Ans
  - Cramm Myrjam, Antwerp
  - Maus Katelijne, Antwerp
  - Debanterlé Stéphane, Barvaux
  - Bourcy Gaelle, Bastogne
  - Deckers Clementine B, Bastogne
  - Vercruysse Klaas, Berchem
  - Balligand Elie, Beringen
  - De Wilde Kristien, Beveren
  - Maes Marc, Beverlo
  - Van De Plas Flip, Boechout
  - Haemels Maria-Magdalena, Boortmeerbeek
  - Cloetens Hanne, Bruges
  - Maryssael Mia, Bruges
  - Freson Micheline, Damme
  - De Meulemeester Marc, Gozée
  - Van Rossem Inès, Halle
  - Compes Annick, Hannut
  - (Mingneau Jannick) Bourguignon Sofie, Heers
  - De Walsche Bram, Herentals
  - Van Immerseel Ilke, Hove
  - Devolder Tyrone, Kortrijk
  - Maertens Katrien, Kortrijk
  - Vanderbauwhede Stefanie, Kortrijk
  - Staelens Toon, Lauwe
  - Van Der Auwera Jolien, Lauwe
  - Marganne Anneline, Liège
  - Lambert Fabienne, Liège
  - Maury Olivier, Linkebeek
  - Saintmar Hélène, Marche-en-Famenne
  - Moeremans Paul, Mechelen
  - Heyvaert Goedele, Merchtem
  - Muylaert Peter, Merelbeke
  - Peetermans Luc, Mol
  - Wuyts Tinne, Mol
  - Pierard Virginie, Monceau-sur-Sambre
  - Grosjean Joël, Mont-sur-Marchienne
  - Andries Laura, Mortsel
  - De Groote Jaron, Oudenaarde
  - Steeno Pieter, Putte
  - Lemiengre Marieke, Roeselare
  - Cardon Philippe, Sambreville
  - Meuris Michel, Spa
  - De Neef Sara, Tienen
  - Op De Beeck Sabine, Turnhout
  - Froidcoeur Xavier, Wanze
  - Tilquin Marlene, Wanze
  - Janssen Reinhilde, Watervliet
  - Bayens Kris, Weelde
  - Klaasen Geert, Weelde
  - Hertegonne Nele, Zottegem

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie the results in our publications will be made available upon request. The IPD set will consist of deidentified participant data. It can be obtained by contacting the research team at KU Leuven: PI, catharina.mathei@kuleuven.be; trial coordinator, marc.vannuland@kuleuven.be; project manager, kristien.coteur@kuleuven.be. Each request before September 2023 will be reviewed by the Sponsor.
  In addition to the IPD set, we will also make the study protocol available through an open access publication, and have registered the trial on clinicaltrials.gov (NCT03937180). The informed consent forms are also publicly available through the trial website (www.bigbirdtrial.com), where the clinical study report will also be disseminated at the end of the trial, after approval of the funder KCE.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: All IPD will be available upon request, after publication of the results concerning the primary outcome, starting six months after publication. The IPD set can be requested until September 2023. For any request later than this date, follow-up by the Sponsor cannot be guaranteed.
Access Criteria: Reuse of the IPD set is only allowed for non-profit research, with correct reference to the original research and Sponsor.

REFERENCES:
- [Derived] Coteur K, Van Nuland M, Schoenmakers B, Anthierens S, Van den Broeck K. Implementing Blended Care to Discontinue Benzodiazepine Receptor Agonist Use for Insomnia: Process Evaluation of a Pragmatic Cluster Randomized Controlled Trial. JMIR Form Res. 2023 Apr 7;7:e43738. doi: 10.2196/43738. PMID 37027198
- [Derived] Coteur K, Henrard G, Schoenmakers B, Laenen A, Van den Broeck K, De Sutter A, Anthierens S, Devroey D, Kacenelenbogen N, Offermans AM, Van Nuland M. Blended care to discontinue benzodiazepine receptor agonists use in patients with chronic insomnia disorder: a pragmatic cluster randomized controlled trial in primary care. Sleep. 2023 Apr 12;46(4):zsac278. doi: 10.1093/sleep/zsac278. PMID 36413221
- [Derived] Coteur K, Van Nuland M, Vanmeerbeek M, Henrard G, Anthierens S, Van den Broeck K, De Sutter A, Creupelandt H, Devroey D, Van Overmeire R, Offermans AM, Kacenelenbogen N, Laenen A, Mathei C. Effectiveness of a blended care programme for the discontinuation of benzodiazepine use for sleeping problems in primary care: study protocol of a cluster randomised trial, the Big Bird trial. BMJ Open. 2020 Feb 18;10(2):e033688. doi: 10.1136/bmjopen-2019-033688. PMID 32075832

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT03937180/Prot_SAP_000.pdf